CLINICAL TRIAL: NCT00032578
Title: CSP #478 (FeAST-DNA), Genetic Tissue Banking in VA Clinical Research: A Cooperative Studies Program Demonstration Project
Brief Title: VA Genetic Tissue Banking
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 478Fe
Record Dates: First submitted 2002-03-27; First posted 2002-03-28 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2006-06

CONDITIONS: Tissue Banking

SUMMARY:
This project is a program-wide genetic tissue databank for the Department of Veterans Affairs Cooperative Studies Program (CSP). The genetic tissue bank has four components: a central repository for DNA and other genetic tissue specimens; a Scientific Advisory Committee of individuals with expertise in the genetics and epidemiology of diseases with special importance to the VA (including cardiovascular, neurologic, respiratory, psychological and other disorders); an Ethics Oversight Committee of individuals with expertise in bioethics and the law, as they apply to the collection and use of genetic tissue, and a Coordinating Center that administers the tissue bank, coordinates the scientific and ethics oversight committees, maintains central access to clinical study data linked to the tissue bank, and provides statistical analysis.

DETAILED DESCRIPTION:
Intervention: No intervention.

Primary Hypothesis: It is feasible and cost-effective to create a CSP-wide facility for banking genetic tissue in CSP studies.

Study Abstract: This is a program-wide genetic tissue databank for the Department of Veterans Affairs Cooperative Studies Program (CSP). The study has five components: a central repository for DNA and other genetic tissue specimens; a Scientific Advisory Committee of individuals with expertise in the genetics and epidemiology of diseases with special importance to the VA (including cardiovascular, neurologic, respiratory, psychological and other disorders); an Ethical Oversight Committee of individuals with expertise in bioethics and the law, as they apply to the collection and use of genetic tissue, A Veteran's Advisory Group, and a Coordinating Center administers the tissue bank, coordinates the three oversight committees, maintains central access to clinical study data linked to the tissue bank, and provides statistical analysis.

ELIGIBILITY:
This DNA Banking substudy piggybacks on VA Cooperative Studies Clinical Trials. All participants who are randomized to selected CSP clinical trials are eligible to participate in the Banking Initiative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Little Rock VAMC, Little Rock, Arkansas
  - VA Palo Alto Health Care System, Palo Alto, California
  - Louisville VAMC, Louisville, Kentucky
  - Durham VA Medical Center, Durham, North Carolina
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - Salt Lake City VA Medical Center, Salt Lake City, Utah
  - White River Junction VAMC, White River Junction, Vermont
  - Madison VA Medical Center, Madison, Wisconsin